CLINICAL TRIAL: NCT06485427
Title: Safety and Efficacy of Selective Intra-Arterial Cooling Infusion Combined With Endovascular Thrombectomy in Acute Ischemic Stroke: A Multicenter, Randomized Controlled, Subject- and Assessor-Blind Clinical Trials
Brief Title: Safety and Efficacy of Selective Intra-Arterial Cooling Infusion Combined With EVT in Acute Ischemic Stroke
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Shen Li, Professor, Beijing Shijitan Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOCUS
Record Dates: First submitted 2024-06-22; First posted 2024-07-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Ischemic Stroke; Hypothermia
MeSH Terms: conditions — Ischemic Stroke; Hypothermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Subjects will receive best medical management (BMM) plus endovascular therapy (EVT) according to the clinical guidelines.
- IA-SCI group (Experimental): Subjects randomized to the IA-SCI group will receive selective intra-arterial cooling infusion plus BMM and EVT.
  Interventions: Procedure: Selective Intra-arterial Cooling Infusion (IA-SCI)

INTERVENTIONS:
Procedure: Selective Intra-arterial Cooling Infusion (IA-SCI) — Pre-recanalization: During the procedure, the micro-catheter is advanced over a micro-guide wire, traveling up through the neck until it reaches beyond the clot. A 50 mL cold 0.9% saline (4 ℃) is infused intro into the ischemic territory at a rate of 10 mL/min via the micro-catheter. This enables the cold solution to infuse into the ischemic territory prior to revascularization.
  Post-recanalization: After recanalization, cold 0.9% saline (4 ℃) is reinfused into the vessel via the catheter at a rate of 22 mL/min for 10 min, repeated twice with a 10-minute interval between infusions.
  Arms: IA-SCI group

SUMMARY:
This is a multicenter, randomized, controlled, subject- and assessor-blinded clinical trial. The research objective is to evaluate the safety and efficacy of selective intra-arterial cooling infusion combined with endovascular therapy in the treatment of acute anterior circulation large vessel occlusion stroke. This trial aims to enroll 258 subjects. Patients assigned to the control group will receive best medical management (BMM) and endovascular therapy (EVT). Those in the selective intra-arterial cooling infusion group (IA-SCI group) will undergo selective intra-arterial cold saline infusion, in addition to BMM and EVT. Subjects will be interviewed face-to-face at randomization, 24±6 hours, 48±6 hours after randomization, 7±2 days/discharge. Telephone interviews/ face-to face interviews will be performed at 30±3 days and 90±7 days after randomization. The primary outcome is the distribution of Modified Rankin Score at 90±7days after randomization.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is the leading cause of death and disability in China. Randomized trials involving patients with acute stroke due to large-artery occlusion in the anterior circulation have shown a benefit of endovascular therapy (EVT). Although EVT achieves successful recanalization in over 80% of patients, only 46% of patients are functionally independent (mRS 0-2) after the intervention . Therefore, new ancillary therapeutic strategies are needed to further improve the clinical outcomes.

Therapeutic systemic hypothermia has been suggested to be one such potential approach offering a viable neuroprotective strategy. However, several adverse events associated with the systematic hypothermia treatment have been reported. Those offset the therapeutic benefits of systemic hypothermia. Selective intra-arterial cooling infusion (IA-SCI) targets precisely the ischemic brain tissue with the infusion of hypothermic solutions. This approach induces a state of mild hypothermia in the ischemic region without causing substantial drops in core body temperature, thereby minimizing the incidence of systemic side effects. Previous studies have shown that IA-SCI with cold saline combined with EVT in AIS is safe and feasible.

Hence, the investigators design a multicenter, randomized, controlled, subject- and assessor-blinded clinical trial. The objective of this trial is to further explore the safety and efficacy of selective intra-arterial cooling infusion combined with EVT in the treatment of acute anterior circulation large vessel occlusion stroke, and 258 subjects will be enrolled. Subjects assigned to the control group will receive best medical management (BMM) and endovascular therapy (EVT). Those in the selective intra-arterial cooling infusion group (IA-SCI group) will undergo selective intra-arterial cold saline infusion, in addition to BMM and EVT. Subjects will be interviewed face-to-face at randomization, 24±6 hours, 48±6 hours after randomization, 7±2 days/discharge. Telephone interviews/ face-to face interviews will be performed at 30±3 days and 90±7 days after randomization. The primary outcome is the distribution of Modified Rankin Score at 90±7days after randomization.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 and ≤ 80.
2. Clinical signs consistent with acute ischemic stroke with large vessel occlusion in the anterior circulation (intracranial segment of the internal carotid artery, middle cerebral artery M1 segment) demonstrated with CTA/MRA/DSA.
3. NIHSS score obtained prior to randomization ≥ 6 and ≤ 25.
4. Modified Rankin Scale ≤ 1 prior to qualifying stroke.
5. Arterial puncture performed within 24 hours from symptom onset or LKW.
6. For the patients with symptom onset within 6 hours, the ASPECT score ≥ 6; for the patients with onset within 6-24 hours, the therapy should meet the imaging criteria of DAWN or DEFUSE-3 trial.
7. Patient/Legally Authorized Representative has signed the Informed Consent Form.

Exclusion Criteria

1. Baseline CT/MRI confirms the presence of multiple vascular territory acute strokes.
2. Baseline CT/MRI confirms the presence of arterial dissection.
3. Evidence of intracranial hemorrhage or hemorrhagic transformation before thrombectomy.
4. Known allergies or intolerances to antiplatelet agents, anticoagulation drugs, iodinated contrast and/or anesthetics.
5. Severe infection (e.g. sepsis) or multiple organ failure.
6. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 3. Patients on factor Xa inhibitor for 48 hours ago must have a normal APTT.
7. Baseline platelet count < 50 × 10^9/L.
8. Blood glucose concentration<50 mg/dL (2.7 mmol/L) or >400 mg/dL (22.2 mmol/L).
9. Refractory hypertension that is difficult to control by medication (Defined as persistent systolic blood pressure>185 mmHg or diastolic blood pressure>110 mmHg).
10. Previous NHYA>1.
11. Untreated moderate or severe coronary artery stenosis, or previous coronary artery bypass surgery.
12. Undergoing hemodialysis or peritoneal dialysis; known severe renal insufficiency with glomerular filtration rate < 30 mL/min or serum creatinine >220 mmol/L (2.5 mg/dL).
13. Known intracranial aneurysm, and cerebral arteriovenous malformation.
14. Malignant brain tumor or CNS infection.
15. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations (e.g., dementia or mental illness)
16. Female who is pregnant or lactating at time of admission.
17. Anticipated life expectancy < 6 months.
18. Current participation in another investigational drug or device study.
19. For other reasons, the responsible clinicians believe that the patient is not suitable for continued treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of Modified Rankin scale | 90 ±7days
  the distribution of Modified Rankin scale (mRS) [ranging from 0 (normal) to 6 (death)]

SECONDARY OUTCOMES:
Percentage of functional independence (mRS scale 0-2) | 90 ±7days
  the percentage of mRS scale 0-2 (Modified Rankin scale [ranging from 0 (normal) to 6 (death)])
Percentage of favorable outcome (mRS scale 0-1) | 90 ±7days
  the percentage of mRS scale 0-1(Modified Rankin scale [ranging from 0 (normal) to 6 (death)])
Final infarction volume | 7±2 days/discharge
  A plain computed tomography (CT) scan will be performed. The infarct area is defined as the low-density area. The infarct area is semi-automatically delineated by the software. The infarct volume= the sum of the infarct area of each layer × layer thickness (5mm).
The changes of infarction volume | 7±2 days/discharge
  the changes of infarction volume between baseline and 7±2 days/discharge assessed by CT
National Institute of Health stroke scale (NIHSS) score | 7±2 days/discharge
  National Institute of Health stroke scale (NIHSS) score [ranging from 0 to 42 points, with higher numbers indicating greater severity]
Barthel Index score | 7±2 days/discharge
  the Barthel Index score [the sum of the score ranging from 0 to 100, with 100 being the most independent level of function]
Rapid neurologic improvement | 24±12 hours
  Rapid neurologic improvement is defined as a reduction of ≥8 on the National Institutes of Health Stroke Scale [ranging from 0 to 42 points, with higher numbers indicating greater severity] or National Institutes of Health Stroke Scale zero to one 24 hours after thrombectomy.
Changes in ipsilateral tympanic membrane temperature | during surgery.
  Changes in ipsilateral tympanic membrane temperature before and after intra-arterial cooling infusion in the IA-SCI group.
Power spectral density (PSD) assessed by continuous electroencephalogram (EEG) | within 7±2 days/discharge
  PSD is estimated using Welch's periodogram from EEG.
(delta+theta)/(alpha+beta) power ratio (DTABR) assessed by continuous electroencephalogram (EEG) | within 7±2 days/discharge
  DTABR is calculated using the absolute power for each of spectral band on EEG.
Delta/alpha power ratio (DAR) assessed by continuous electroencephalogram (EEG) | within 7±2 days/discharge
  DAR is calculated using the absolute power for each of spectral band on EEG.
Brain symmetry index (BSI) assessed by continuous electroencephalogram (EEG) | within 7±2 days/discharge
  BSI is calculated using the power values from both left and right hemispheres from EEG.
Symptomatic intracranial hemorrhage | 24±12 hours
  Defined as any intracranial hemorrhage accompanied by neurological deterioration (NIHSS score increased by more than 4 points compared with the lowest NIHSS score at enrollment or during hospitalization) or death caused by any cerebral hemorrhage according to the ECASS III study.
Any intracranial hemorrhage | 24±12 hours
  any intracranial hemorrhage assessed by CT
Intracranial arterial vasospasm after IA-SCI that requires further therapeutic intervention. | during operation
  Patients with vasospasm confirmed by DSA and requiring further therapeutic intervention
Proportion of subjects with pulmonary, urinary tract infection and gastroenteritis | 7±2 days/discharge
  the proportion of patients with pulmonary, urinary tract infection and gastroenteritis according to the Centers for Disease Control and Prevention (CDC)/ National Healthcare Safety Network (NHSN) criteria.
Proportion of subjects with coagulation abnormalities | 24±12 hours
  Defined as abnormal coagulation function
Proportion of subjects with electrolyte imbalance | 24±12 hours
  Defined as any abnormal findings, including hypernatremia, hyponatremia, hyperkalemia, or hypokalemia.
Changes in core temperature before and after intra-arterial cooling infusion in the IA-SCI group. | During operation
  Changes in rectal temperature before and after intra-arterial cooling infusion in the IA-SCI group.
any death | 90±7 days
  any death
other AE/SAE | 90±7 days
  other adverse events/ serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shen Li, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (9):
- China (9):
  - The Second Hospital and Clinical Medical School, Lanzhou University, Lanzhou, Gansu
  - Department of Neurosurgery, Nanshi Hospital of Nanyang, Nanyang, Henan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Peking University Internation Hospital, Beijing
  - 967 Hospital of the Joint Logistics Support Force of PLA, Dalian
  - Dalian Municipal Central Hospital, Dalian
  - The First Affiliated Hospital of Harbin Medical University, Ha’erbin
  - Affiliated Hospital of Inner Mongolia University for the Nationalities, Tongliao

IPD SHARING:
Plan to Share IPD: No